CLINICAL TRIAL: NCT06615440
Title: Management and Outcome of Scorpion Sting in Children
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mahmoud Hamdy Abdelaziz Sayed, Doctor, Assiut University
Other Study IDs: Management of scorpion sting
Record Dates: First submitted 2024-09-16; First posted 2024-09-26 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Scorpion Stings
MeSH Terms: conditions — Scorpion Stings | interventions — Adrenergic alpha-Antagonists

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Alpha blocker — prazosin will be given to all children with systemic manifestations (orally or by nasogastric tube) at a dose of 30 μg/kg/dose;first repeat dose at 3 h followed by every 6 h till recovery. All patients will be monitored for clinical improvement with vital signs

SUMMARY:
To determine the clinical characteristics of children with scorpion sting and implement guidelines for management of those children and observe the outcome

DETAILED DESCRIPTION:
Scorpion envenomation is a severe,sometimes fatal medical condition especially in children .Worldwide,there are more than 1.2 million scorpion stings each year,mostly in tropical and subtropical regions.Every year,more than 420,000 snake bite,scorpion sting and spider bite incidents occur in the Middle East and North Africa (MENA).In the region of Assiut,in the South of Egypt,the annual incidence and mortality by scorpion stings has been reported to be 88 and 5.5 per 100,000 inhabitants.There are 1500 sub species of scorpions in the globe,and 50 of those have venom that is harmful to humans.The most toxic scorpion families are the Buthidae family.The MENA region is home to 27 species of scorpions from three families:theButhidae,Hemiscorpiidae,and Scorpionidae.Significant morbidity and mortality are caused by scorpion stings .In addition to local effectslikeredness,pain,burning,and swelling,scorpion venom exhibits variability among sub species and has a complex structure made up of neurotoxic proteins,salts,acidic proteins,and organic compounds.These components can cause neurological,cardiovascular,hematologic,and renal side effects.Because scorpion venoms are complex mixtures of several toxins,including cardiotoxins,nephrotoxins,hemolytictoxins,and neurotoxins,there is a possible danger of developing severe and frequently deadly clinical consequences.Heart failure and pulmonary edema are the main causes of mortality .As regards management of scorpion sting early antivenom treatment is recommended but its value remains controversial as it may cause anaphylactic reactions .Furthermore the majority of cases need supportive treatment to alleviate the cardiovascular effect.Cardiovascular symptoms respond well to vasodilators such as alpha-1blockers like prazosin.Prazosinis considered a physiological and pharmacological antidote to scorpion venom action.It antagonizes the after-effects of venom-liberated catecholamines.Since the use of prazosin with antivenom the recovery from scorpion sting has been hastened and mortality rate has been reduced from 30% to 1%.Uptill now there are no guidlines implemented at our hospital for the management of scorpion sting so that our study will aim at implementing guidelines for management of children with scorpion sting and observe the outcome of those children.The guidelines used are those recommended from the Egyptian ministry of health and Population with the addition of prazosin as many studies have concluded the benefits of prazosin

ELIGIBILITY:
Inclusion Criteria:

- All children under 18 years with definite history of scorpion sting

Exclusion Criteria:

* Children with no definite history of sting or more than 18 years

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Prazosin will be given to all children with systemic manifestations (orally or by nasogastric tube) at a dose of 30 μg/kg/dose;first repeat dose at 3 h followed by every 6 h till recovery.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2024-11 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Role of prazosin in management of scorpion sting | Baseline
  Prazosin, a post synaptic alpha blocker, can be recommended as an effective drug in the treatment of serious scorpion enve- nomations with significant sympathetic symptoms.antagonises the effects of catecholamines thereby preventing further damage of myocardium though it cannot reverse the damage
  Prazosin will be given to all children with systemic manifestations (orally or by nasogastric tube) at a dose of 30 μg/kg/dose;first repeat dose at 3 h followed by every 6 h till recovery.To determine the clinical characteristics of children with scorpion sting and implement guidelines for management of those children and observe the outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Children hospital Assiut University, Asyut, Egypt

REFERENCES:
- [Background] WorldHealthOrganization.WHOExpertCommitteeonBiologicalStandardization, sixty-seventhreport.Licence:CCBY-NC-SA3.0IGO.Geneva;2017.Available: https://www.who.int/publications/i/item/9789241210133
- [Background] Rajniti Prasad et al. Indian J Pediatr. 2011 May.https://link.springer.com/article/10.1007/s12098-010-0265-0
- [Background] Kumar,Rakesh.AnupdateonepidemiologyandmanagementpracticesofScorpio nenvenomationinIndia.*JournalofFamilyMedicineandPrimaryCare*.11(9),493 2- 4935,September2022.DOI:10.4103/jfmpc.jfmpc_2300_2
- [Background] Mohamad IL, Elsayh KI, Mohammad HA, Saad K, Zahran AM, Abdallah AM, Tawfeek MS, Monazea EM. Clinical characteristics and outcome of children stung by scorpion. Eur J Pediatr. 2014 Jun;173(6):815-8. doi: 10.1007/s00431-013-2244-8. Epub 2014 Jan 3. PMID 24384790
- [Background] FarghalyWM,AliFA(1999)Aclinicalandneurophysiologicalstudyofscorpion envenomationinAssiut,UpperEgypt.ActaPaediatr88(3):290-294.
- [Background] Bawaskar HS, Bawaskar PH. Clinical profile of severe scorpion envenomation in children at rural setting. Indian Pediatr. 2003 Nov;40(11):1072-5. PMID 14660839
- [Background] https://scholar.google.com/scholar_lookup?journal=Int.+J.+Bioinform.+Biomed.+Eng.&amp;amp;amp;title=Scorpion+sting+in+different+regions+of+Sudan:+epidemiological+and+clinical+survey+among+university+students&amp;amp;amp;author=N.+Ali&amp;amp;amp;author=N.+O+M+Ali&amp;amp;amp;publication_year=2015&amp;amp;amp;